CLINICAL TRIAL: NCT05911360
Title: A Phase 3b, Multicenter, Single-arm, Open-label Study Evaluating the Efficacy, Safety, and Tolerability of Switching to DTG/3TC Single Tablet Regimen Administered Once Daily From a Bictegravir/Emtricitabine/Tenofovir Alafenamide Single Tablet Regimen in People Living With HIV of at Least 50 Years of Age Who Are Virologically Suppressed
Brief Title: A Study to Evaluate Efficacy, Safety and Tolerability in Antiretroviral Therapy (ART)-Experienced Participants of at Least 50 Years of Age Living With Human Immunodeficiency Virus (HIV) With Virologic Suppression Who Switch to DTG/3TC FDC From BIC/FTC/TAF
Acronym: EYEWITNESS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 219516; 2022-503137-66-00 (Other: EU CT number)
Record Dates: First submitted 2023-06-09; First posted 2023-06-22 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: HIV; HIV Infections
Keywords: Human Immunodeficiency Virus (HIV)-1; Dolutegravir; Lamivudine; Bictegravir; Emtricitabine; Tenofovir alafenamide; Dovato; Biktarvy; Switch study; ≥ 50 years
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants Receiving DTG/3TC FDC (Experimental)
  Interventions: Drug: DTG/3TC

INTERVENTIONS:
Drug: DTG/3TC — DTG/3TC FDC will be administered once daily.

SUMMARY:
The study aims at evaluating the maintenance of virologic suppression of dolutegravir/lamivudine (DTG/3TC) fixed dose combination (FDC) at Week 48 post-switch from bictegravir/emtricitabine/tenofovir alafenamide (BIC/FTC/TAF) in participants living with Human Immunodeficiency Virus Type 1 (HIV-1) who are of at least 50 years of age and above.

ELIGIBILITY:
Inclusion Criteria:

* Participants living with HIV-1 with documented plasma HIV-1 RNA <50 c/mL within 3 months prior to Screening.
* Participants must have been on uninterrupted antiretroviral therapy (ART) for ≥1 year (except for brief periods [less than 30 days] where all ART was stopped due to tolerability and/or safety concerns).
* Participants must be on uninterrupted BIC/FTC/TAF for at least 6 months prior to Screening.
* Participants with plasma HIV-1 RNA <50 c/mL at Screening.
* Participants with no known prior regimen switches due to documented virologic failure (defined as a confirmed plasma HIV 1 RNA ≥200 c/mL).
* Participants with unknown full treatment/clinical history beyond 5 years prior to Screening may be eligible upon discussion and agreement with the medical monitor.

Exclusion Criteria:

* Women participants who are pregnant or breastfeeding or plan to become pregnant or breastfeed during the study.
* Participants with any evidence of an active Centers for Disease Control and Prevention (CDC) Stage 3 disease, EXCEPT cutaneous Kaposi's sarcoma not requiring systemic therapy. Historical or current CD4 cell counts less than 200 cells/cubic millimetre (mm^3) are not exclusionary.
* Participants with signs and symptoms which, in the opinion of the Investigator, are suggestive of active severe acute respiratory syndrome-related coronavirus (SARS-CoV-2) infection within 14 days prior to enrolment.
* Participants with severe hepatic impairment (Class C) as determined by Child-Pugh classification.
* Evidence of hepatitis B virus (HBV) infection based on the results of testing at Screening for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (anti-HBc), hepatitis B surface antibody (anti-HBs) and HBV deoxyribonucleic acid (DNA) as follows:

  1. Participants positive for HBsAg are excluded;
  2. Participants negative for anti-HBs but positive for anti-HBc (negative HBsAg status), whether negative or positive for HBV DNA, are excluded;
  3. Participants positive for anti-HBc (negative HBsAg status) and positive for anti-HBs (past and/or current evidence) are immune to HBV and are not excluded.
* Participants with unstable liver disease (as defined by any of the following: presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice or cirrhosis), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment).
* Participants with history of liver cirrhosis with or without hepatitis viral co-infection.
* Participants with untreated syphilis infection (positive rapid plasma reagin [RPR] at Screening without clear documentation of treatment). Participants who are at least 7 days post completed treatment are eligible.
* Participants with history or presence of allergy or intolerance to the study treatment or their components or drugs of their class or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical, anal or penile intraepithelial neoplasia.
* Participants who in the investigator's judgment, poses a significant suicidality risk. Participant's history of suicidal behavior and/or suicidal ideation should be considered when evaluating for suicide risk.
* Participants with any evidence of any major 3TC resistance associated mutations (M184V/I and/or K65R and/or MDR) or presence of any major Integrase strand transfer inhibitor (INSTI) resistance associated mutation in any available prior resistance genotype assay test result. All available historical resistance reports with HIV-1 reverse transcriptase or integrase genotypic data must be provided to ViiV after screening and before enrollment for review by ViiV Virology.
* Participants with any verified Grade 4 laboratory abnormality with the exception of Grade 4 lipid abnormalities.
* Alanine aminotransferase (ALT) ≥5 times the upper limit of normal (ULN) or ALT ≥3xULN and bilirubin ≥1.5xULN (with greater than [>]35 percentage [%] direct bilirubin).
* Participant has estimated creatine clearance <30 millilitres per minute (mL/min) per 1.73 square meter (m^2) using the refitted, race-neutral Chronic Kidney Disease Epidemiology Collaboration (CKD-EPIcr_R) method.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2026-01-13 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Plasma HIV-1 Ribonucleic Acid (RNA) Greater Than or Equal to (≥)50 Copies/Millilitre (c/mL) per Snapshot Algorithm at Week 48 | Week 48

SECONDARY OUTCOMES:
Number of Participants With Plasma HIV-1 RNA ≥50 c/mL per Snapshot Algorithm at 24 and 96 Weeks | Weeks 24 and 96
Number of Participants With Plasma HIV-1 RNA Less Than (<)50 c/mL per Snapshot Algorithm at 24, 48 and 96 Weeks | Weeks 24,48, and 96
Absolute Values for Cluster of Differentiation 4 (CD4+) Cells Count at 24, 48 and 96 Weeks | Weeks 24,48, and 96
Change From Baseline in CD4+ Cells Count at 24, 48 and 96 Weeks | Baseline (Day 1) and at Weeks 24,48, and 96
Absolute Values for CD4: Cluster of Differentiation 8 (CD8) Ratio at 24, 48 and 96 Weeks | Weeks 24,48, and 96
Change From Baseline in CD4:CD8 Ratio at 24, 48 and 96 Weeks | Baseline (Day 1) and at Weeks 24,48, and 96
Number of Participants With Disease Progression Through Weeks 24, 48 and 96 | Weeks 24, 48, and 96
Number of Participants who Meet Confirmed Virologic Withdrawn Criterion With Viral Resistance Over Time | Up to Week 96
Number of Participants With Treatment Related Non-serious Adverse Events, all Serious Adverse Events (SAEs), and AEs Leading to Treatment Discontinuation | Up to Week 96
  A treatment related AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, and considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations judged by physician, is associated with liver injury and impaired liver function.

CONTACTS AND LOCATIONS:
Locations (53):
- United States (24):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Palm Springs, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Berkley, Michigan
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Austin, Texas
- Austria (2):
  - GSK Investigational Site, Innsbruck
  - GSK Investigational Site, Vienna
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
- Canada (2):
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (3):
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Orléans
  - GSK Investigational Site, Paris
- Germany (3):
  - GSK Investigational Site, Freiburg im Breisgau
  - GSK Investigational Site, Hanover
  - GSK Investigational Site, München
- Italy (4):
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Modena
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Torino
- Mexico (2):
  - GSK Investigational Site, Mérida
  - GSK Investigational Site, Monterrey
- Netherlands (3):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Utrecht
- Portugal (2):
  - GSK Investigational Site, Porto
  - GSK Investigational Site, Vila Nova de Gaia
- Spain (4):
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Manresa Barcelona
  - GSK Investigational Site, Sabadell Barcelona
  - GSK Investigational Site, Zaragoza
- United Kingdom (2):
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/